CLINICAL TRIAL: NCT07354893
Title: Evaluation of an Educational Intervention on Knowledge and Awareness of Infectious Risk in Splenectomized Patients and on Their Satisfaction With Vaccination Management in an Intra-hospital Outpatient Setting.
Brief Title: Evaluation of the Effectiveness of an Educational Intervention in Splenectomized Patients
Acronym: SPLE-VAC
Status: Recruiting | Type: Observational
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Laurenti Patrizia, Professor, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Other Study IDs: 8123
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Splenectomized Patients; Splenectomy; Splenectomy; Status; Asplenia
Keywords: OPSI; infection risk; Infection Prevention; Preventive measures; Vaccination; asplenia; splenectomy; splenectomized patients; post splenectomy infections

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Educational intervention for asplenic patients — an educational intervention aimed at informing patients about the condition of asplenia, the associated infectious risks, and the main preventive measures, with particular emphasis on vaccination prophylaxis. To support the intervention, educational materials will be distributed, including an informational brochure and the "Recommended Vaccinations for Asplenic Patients" schedule.

SUMMARY:
The absence or dysfunction of the spleen is associated with a substantially increased risk of invasive infections that may rapidly progress to fulminant sepsis, including overwhelming post-splenectomy infection (OPSI), a medical emergency with high mortality. Although the risk is greatest in the first two years after splenectomy, it persists lifelong. Preventing infections in patients with anatomical or functional asplenia requires an integrated strategy that includes patient education, early recognition of symptoms, behavioral measures, antibiotic prophylaxis when indicated, and vaccination.

Post-splenectomy immunization has been shown to reduce OPSI incidence. Regional and international guidelines recommend vaccination against pneumococcus, Haemophilus influenzae type b, meningococcus (B and ACWY), herpes zoster, diphtheria-tetanus-pertussis, measles-mumps-rubella-varicella, and annual influenza. However, adherence to these recommendations is frequently suboptimal, often due to limited awareness among patients and healthcare professionals.

This study involves the intra-hospital vaccination team providing structured vaccination consultations to splenectomized patients hospitalized at the Fondazione Policlinico Universitario "A. Gemelli" IRCCS. During ward consultations, patients receive an educational intervention on asplenia-related infectious risks and preventive measures, supported by standardized informational materials. Effectiveness is evaluated using a pre-post questionnaire assessing knowledge and awareness. Patients completing the vaccination pathway at the outpatient clinic also complete a questionnaire assessing their experience with vaccination management in an intra-hospital setting.

DETAILED DESCRIPTION:
This is a prospective, observational patient registry conducted at a single academic hospital. Adult patients undergoing splenectomy at the Fondazione Policlinico Universitario A. Gemelli IRCCS are consecutively identified through routine inpatient clinical workflows and enrolled after written informed consent.

Clinical, sociodemographic, and vaccination-related data are collected as part of standard care by the intra-hospital vaccination clinic and recorded in a dedicated database using predefined variables. Patient-reported outcomes are assessed using structured questionnaires administered before and after an educational intervention and, for patients completing the vaccination pathway, at the end of follow-up.

The registry allows longitudinal follow-up to monitor patient education, vaccination uptake, completion of recommended schedules, and post-discharge continuity of care. Follow-up data are collected during outpatient visits or, when necessary, via structured telephone interviews.

Data quality is ensured through standardized data collection procedures, use of validated questionnaires, and cross-verification of vaccination data using independent institutional sources. All data are pseudonymized and managed in compliance with applicable data protection regulations. The study is conducted according to Good Clinical Practice, Good Epidemiological Practice, and the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years old)
* Patients splenectomized at FPG for whom a vaccination consultation is requested during hospitalization
* Patients who provide signed informed consent to participate in the study and for the processing of personal data for research purposes

Exclusion Criteria:

* Minor patients
* Lack of signed informed consent for participation in the study and for the processing of personal data for research purposes
* Patients splenectomized at other healthcare facilities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients splenectomized at the Fondazione Policlinico Universitario A. Gemelli IRCCS, identified during consultation activities in the requesting wards and/or managed by the hospital outpatient vaccination clinic for frail patients.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-01-13 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-01-13 (Estimated)

PRIMARY OUTCOMES:
Change in Infectious Risk Knowledge, Vaccination Attitudes, and Risk Perception Score | 24 months
  Change from baseline to post-intervention in patients' knowledge of infectious risk, attitudes toward vaccination, and perception of infectious risk following an educational and counseling intervention. The outcome is assessed in splenectomized patients identified and/or managed by the intra-hospital outpatient clinic of the Fondazione Policlinico Universitario "A. Gemelli" IRCCS (FPG).
  Measure Description:
  Infectious Risk and Vaccination Awareness Questionnaire for Splenectomized Patients (specifically developed and validated questionnaire). The total score ranges from 16 to 80, with higher scores indicating greater knowledge, more favorable attitudes toward vaccination, and higher perceived infectious risk.

SECONDARY OUTCOMES:
Patient Experience with Vaccination Prophylaxis Management Score | 24 months
  Patient experience related to the management of vaccination prophylaxis in an intra-hospital outpatient setting, assessed during follow-up outpatient visits.
  Measure Description:
  Patient Experience with Vaccination Prophylaxis Questionnaire (validated questionnaire derived from the literature). The total score ranges from 13 to 65, with higher scores indicating a more positive patient experience.
Association Between Infectious Risk Knowledge Score and Socio-demographic Characteristics | 24 months
  Correlation between patients' infectious risk knowledge and awareness levels and socio-demographic characteristics (e.g., age, sex, educational level, clinical characteristics), aimed at identifying factors useful for the personalization of educational interventions.
  Measure Description:
  Infectious Risk and Vaccination Awareness Questionnaire for Splenectomized Patients. Associations will be evaluated using correlation coefficients and regression parameters.
Adherence to the Intra-hospital Vaccination Pathway | 24 months
  Adherence to the intra-hospital vaccination pathway among splenectomized patients managed by the outpatient clinic, including enrollment in the pathway and administration of recommended vaccinations.
  Measure Description:
  Proportion (expressed in percentage, %) of patients enrolled in the vaccination pathway and proportion of recommended vaccinations administered per patient. Values range from 0% to 100%, with higher percentages indicating greater adherence.

CONTACTS AND LOCATIONS:
Overall Officials: LAURENTI PATRIZIA, PROFESSOR, Principal Investigator — Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Locations (2):
- Italy (2):
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Rome, Lazio
  - Fondazione Policlinico Universitario A. Gemelli IRCCS, Roma

IPD SHARING:
Plan to Share IPD: Undecided